CLINICAL TRIAL: NCT06822777
Title: A Randomized Controlled Trial of RISE for Nurse Preceptors
Brief Title: RISE for Nurse Preceptors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2251716
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-07

CONDITIONS: Mental Health; Resilience; Self-Compassion; Empowerment; Well-Being, Psychological; Burnout, Healthcare Workers
MeSH Terms: conditions — Psychological Well-Being; Empowerment; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intervention group will attend the RISE for Nurse Preceptors program, which consists of nine 90-minute weekly psychoeducational group sessions facilitated by a licensed mental health counselor (LMHC)
  Interventions: Behavioral: RISE for Nurse Preceptors Program
- Wait-list control group (Active Comparator): Control group will attend the RISE for Nurse Preceptors program after the 6-month wait-list period
  Interventions: Behavioral: RISE for Nurse Preceptors Program

INTERVENTIONS:
Behavioral: RISE for Nurse Preceptors Program — Psychoeducational group program designed to impact resilience, insight, self-compassion, and empowerment

SUMMARY:
The purpose of this study is to determine whether RISE for Nurse Preceptors has a significant impact on nurse preceptors' burnout, resilience, insight, self-compassion, and empowerment, as well as mental well-being, in their personal lives and their working environment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old
2. Licensed as an RN
3. Employed by AdventHealth Rocky Mountain Region
4. Completion of the AdventHealth preceptor training
5. Has precepted ≥ 48 hours within the past calendar year in an AdventHealth hospital setting or outpatient emergency center
6. Able to speak, read, and understand English fluently
7. Able to provide informed consent
8. Willing and able to comply with all study procedures and requirements for the duration of the study.

Exclusion Criteria:

1. Has precepted < 48 hours within the past calendar year
2. Does not pass the brief risk assessment in the pre-intervention introduction meeting with the LMHC facilitator
3. Unwilling or unable to comply with all study procedures and requirements for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Professional Quality of Life Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  30-item questionnaire with the following response categories: 1=never, 2=rarely, 3=sometimes, 4=often, 5=very often

SECONDARY OUTCOMES:
Posttraumatic Growth Inventory | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  21-item questionnaire with a scale of 0-5, with 0 meaning I did not experience this change as a result of my crisis; and 5 meaning I experienced this change to a very great degree as a result of my crisis
Brief Resilience Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  6-item questionnaire with the following response categories: 1=strongly agree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree
Self-Reflection and Insight Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  20-item questionnaire with a scale of 1-6; with 1 meaning strongly disagree; and 6 meaning strongly agree
Self-Compassion Scale - Short Form | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  12-item questionnaire with the following response categories: 1=almost never, 2, 3, 4, 5=almost always
Psychological Empowerment Instrument | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  12-item questionnaire with a scale of A-G, with A meaning very strongly disagree; and G meaning very strongly agree
General Self-Efficacy Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  10-item questionnaire with the following response categories: 1=not at all true, 2=barely true, 3=moderately true, 4=exactly true
Perceived Stress Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  10-item questionnaire with the following response categories: 0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often
Moral Injury Outcomes Scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  14-item questionnaire with the following response categories: 0=strongly agree, 1=disagree, 2=neither agree or disagree, 3=agree, 4=strongly agree
Brief COPE | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  28-item questionnaire with a scale of 1-4, with 1 meaning I haven't been doing this at all; and 4 meaning I've been doing this a lot
Generalized Anxiety Disorder - 2 item scale | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  2-item questionnaire with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day
Patient Health Questionnaire - 2 item | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  2-item scale with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day
Preceptor Self-Assessment Tool | Baseline, endpoint, and 1-, 3-, and 6-month follow-up
  40-item scale with the following response categories: 1 (lowest), 2 (low), 3 (average), 4 (high), 5 (highest).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey AK, Sawyer AT, Robinson PS. A Psychoeducational Group Intervention for Nurses: Rationale, Theoretical Framework, and Development. J Am Psychiatr Nurses Assoc. 2023 May-Jun;29(3):232-240. doi: 10.1177/10783903211001116. Epub 2021 Jun 22. PMID 34154451
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Grant, A. M., Franklin, J., & Langford, P. (2002). The Self-Reflection and Insight Scale: A new measure of private self-consciousness. Social Behavior and Personality, 30(8), 821-836.
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] L'Ecuyer K, Subramaniam DS, Reansing C, DuBois JC. Psychometric Testing of the Preceptor Self-Assessment Tool (PSAT)-40 for Nursing Preceptors. J Contin Educ Nurs. 2022 Nov;53(11):491-499. doi: 10.3928/00220124-20221006-06. Epub 2022 Nov 1. PMID 36318709
- [Background] Litz BT, Plouffe RA, Nazarov A, Murphy D, Phelps A, Coady A, Houle SA, Dell L, Frankfurt S, Zerach G, Levi-Belz Y; Moral Injury Outcome Scale Consortium. Defining and Assessing the Syndrome of Moral Injury: Initial Findings of the Moral Injury Outcome Scale Consortium. Front Psychiatry. 2022 Jul 5;13:923928. doi: 10.3389/fpsyt.2022.923928. eCollection 2022. PMID 35873252
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Sawyer AT, Bailey AK, Green JF, Sun J, Robinson PS. Resilience, Insight, Self-Compassion, and Empowerment (RISE): A Randomized Controlled Trial of a Psychoeducational Group Program for Nurses. J Am Psychiatr Nurses Assoc. 2023 Jul-Aug;29(4):314-327. doi: 10.1177/10783903211033338. Epub 2021 Jul 23. PMID 34293934
- [Background] Sawyer AT, Tao H, Bailey AK. The Impact of a Psychoeducational Group Program on the Mental Well-Being of Unit-Based Nurse Leaders: A Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Jun 2;20(11):6035. doi: 10.3390/ijerph20116035. PMID 37297639
- [Background] Sawyer AT, McManus K, Bailey AK. A mixed-methods pilot study of a psychoeducational group programme for nurse managers during the COVID-19 pandemic. J Nurs Manag. 2022 Nov;30(8):4126-4137. doi: 10.1111/jonm.13881. Epub 2022 Nov 13. PMID 36326077
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spreitzer, G. M. (1995). Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal, 38(5), 1442-1465.
- [Background] Stamm, B. H. (2009). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL). http://www.proqol.org.
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649